CLINICAL TRIAL: NCT05746884
Title: Haemostatic Gel Prophylaxis for Post Duodenal Endoscopic Resection Bleeding
Acronym: PURASTAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A02660-43
Record Dates: First submitted 2023-02-13; First posted 2023-02-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Duodenal Bleeding

STUDY DESIGN:
Intervention Model Description: Single-blind, controlled, comparative, randomized, multicentre, international post-marketing follow-up study of a CE marked medical device.
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group with PuraStat® (Experimental): Endoscopic mucosectomy or endoscopic ampullectomy with standard resection technique, per-procedure hemostasis at operator discretion and application of PuraStat®
  Interventions: Procedure: duodenal mucosectomy; Procedure: ampullectomy
- Control Group (Active Comparator): Endoscopic mucosectomy or endoscopic ampullectomy with standard resection technique, per-procedural hemostasis at operator discretion
  Interventions: Procedure: duodenal mucosectomy; Procedure: ampullectomy

INTERVENTIONS:
Procedure: duodenal mucosectomy — Standard resection technique will be performed for duodenal mucosectomy, as well as the usual hemostasis at the discretion of the operator.
Procedure: ampullectomy — Standard resection technique will be performed for ampullectomy, as well as the usual hemostasis at the discretion of the operator.

SUMMARY:
The purpose of this study is to test whether prophylactic application of haemostatic gel will reduce the rate of clinically significant bleeding requiring intervention (such as blood transfusion, admission to hospital, other blood products) following endoscopic resection of advanced duodenal neoplasia compared to standard therapy.

DETAILED DESCRIPTION:
This is a post-marketing follow-up study of a CE marked medical device, controlled, comparative, randomized, multicentre, international single-blind.

The main objective is to evaluate the efficacy and safety of PuraStat in duodenal endoscopic mucosal resection or ampullectomy.

This study will be carried out in France in 3 investigative centers. The duration of patient participation in the study is approximately 37 days depending on the time between the selection and the endoscopic intervention.

ELIGIBILITY:
Inclusion Criteria:

Ampullary lesions

* Single ampullary lesion ≥ 10mm
* Resection via hot ampullectomy, injection/Endoscopic mucosal resection of adjacent lateral spreading component Duodenal Lesions
* ≤ 2 lesions
* Lesion ≥15mm
* Resection via hot Endoscopic mucosal resection
* Morphology: 0-Is, 0-IIa/b/c or combination, submucosal lesions

Exclusion Criteria:

* Inability to provide informed consent (including people with cognitive impairment);
* Pregnant or breastfeeding women;
* Allergy to PuraStat®;
* "Cold" mucosal endoscopic resection;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty;
* Participating patient, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Bleeding rate requiring further intervention within 30 days | 30 days
  Rate of clinically significant delayed postoperative bleeding requiring further intervention within 30 days (such as blood transfusion, packed cell transfusion or administration of other blood products, hospitalization or repeat endoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No